CLINICAL TRIAL: NCT03387033
Title: Role of Virtual Reality (VR) in Decreasing Pain and Anxiety in Patients With Sickle Cell Disease (SCD)
Brief Title: Role of Virtual Reality (VR) in Patients With Sickle Cell Disease (SCD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment closed due to lack of funding
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00082388
Record Dates: First submitted 2017-06-14; First posted 2017-12-29 (Actual); Results first posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Sickle Cell Disease; Virtual Reality; Anxiety; Depression; Cancer
MeSH Terms: conditions — Anemia, Sickle Cell; Anxiety Disorders; Depression; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- VR intervention session (Experimental): The patients will give a pain score as well as fill out GAD-7 and PHQ-9 scores initially. The VR intervention session consists of relaxation narration WITH Virtual Reality session for 20 minutes while wearing the VR device. They will then be again asked to give a pain score and fill out GAD-7, PHQ-9, and PGIC.
  Interventions: Device: Relaxation response and virtual reality (VR) session

INTERVENTIONS:
Device: Relaxation response and virtual reality (VR) session — A 10-minute relaxation response (mindfulness and deep breathing) followed by 10-minute immersive VR session.
  Other Names: NeuTab VR Headset; Mindfulness; Deep breathing; Dynamic Virtual Viewer

SUMMARY:
Patients with sickle cell disease (SCD) and cancer often have complicated courses while hospitalized and often deal with pain, anxiety and depression. Advances in the field of technology provide potential avenues for innovative and improved care models for our patients. Virtual reality (VR) has been recently utilized to improve anxiety and pain in a variety of patient populations including children undergoing elective surgery and children experiencing intravenous cannulation in the Emergency Department. Patients with SCD and cancer, both adults and children, are a group of patients that can benefit from VR as part of their care. Over the past four years, our team has successfully implemented several self-developed mobile applications ("apps") for our patients, in addition to integrating objective data (heart rate, activity, stress) from wearable activity trackers. The investigators now propose implementing a feasibility study followed by a pilot study and randomized-controlled trial of the use of VR in patients with SCD and cancer. The investigators plan to assess pain and anxiety prior to the session as well as following the session in hospitalized patients and outpatients with SCD and cancer. The sessions will include a ten-minute relaxation response introductory narrative segment (deep breathing and mindfulness) followed by a ten-minute narrated and immersive VR. Heart rate will be tracked using an Apple iWatch for 30 minutes prior to the session, during the session, and following the session. We anticipate VR will not only be a feasible method to provide non-pharmacologic treatment, but will also significantly reduce pain and anxiety.

DETAILED DESCRIPTION:
The investigators will perform a feasibility and pilot study evaluating relaxation response (narration leading through deep-breathing, mindfulness, and other relaxation techniques) followed by VR in patients with sickle cell disease (SCD) and caner. The VR headset (NeuTab VR Virtual Reality Headset, Dynamic Virtual Viewer, or similar device) used will be compatible with an iPhone purchased by the PI. The VR session will be narrated by Jon Seskevich, RN. Patients will be provided with a second iPhone to play the recording while the other iPhone is used to display the VR session.

The patients will first be provided a consent form and consented. They will have the opportunity to ask questions prior to and following consent. They will subsequently give a pain score and fill out a GAD-7 (Generalized Anxiety Disorder) and PHQ-9 (Patient Health Questionnaire) form. They will be taught how to use the VR headset. Patients will listen to a recording by Jon Seskevich, RN of a ten-minute relaxation response. An iPhone will then be placed in the VR headset, the recording started, and the headset placed on the patient. The VR scene is available through Provata VR app and has been previously chosen prior to the start of the study. Following this, patients will again give a pain score as well as complete another GAD-7, PHQ-9, Presence Questionnaire, and Patient's Global Impression of Change (PGIC) form. Patients will be asked to fill out pain score and general health questions via the TRU-Pain app. Patients will then be able to ask questions/provide further feedback.

ELIGIBILITY:
Inclusion Criteria:

* These patients must have a diagnosis of chronic or acute pain (current pain or baseline pain score >0) AND
* These patients must have anxiety and depressive symptoms as measured by the GAD-7 or PHQ-9 questionnaires

Exclusion Criteria:

* Patients <8 years old

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nirmish Shah, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
Currently have collaborators at Pitt interested and may expand study pending feasibility and pilot study results.

REFERENCES:
- [Background] Chow CH, Van Lieshout RJ, Schmidt LA, Dobson KG, Buckley N. Systematic Review: Audiovisual Interventions for Reducing Preoperative Anxiety in Children Undergoing Elective Surgery. J Pediatr Psychol. 2016 Mar;41(2):182-203. doi: 10.1093/jpepsy/jsv094. Epub 2015 Oct 17. PMID 26476281
- [Background] Jonassaint CR, Shah N, Jonassaint J, De Castro L. Usability and Feasibility of an mHealth Intervention for Monitoring and Managing Pain Symptoms in Sickle Cell Disease: The Sickle Cell Disease Mobile Application to Record Symptoms via Technology (SMART). Hemoglobin. 2015;39(3):162-8. doi: 10.3109/03630269.2015.1025141. Epub 2015 Apr 1. PMID 25831427
- [Background] Shah N, Jonassaint J, De Castro L. Patients welcome the Sickle Cell Disease Mobile Application to Record Symptoms via Technology (SMART). Hemoglobin. 2014;38(2):99-103. doi: 10.3109/03630269.2014.880716. Epub 2014 Feb 10. PMID 24512633
- See also: National Center for Health Statistics: Mental Health. CDC — https://www.cdc.gov/nchs/fastats/mental-health.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 20 patients were enrolled into the study from the outpatient sickle cell clinic (15%), inpatient unit (15%) and sickle cell day hospital (70%).
Period: Overall Study
Arm/Group | VR Intervention Session
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VR Intervention Session
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 28.5 [19 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Sickle Cell Disease (SCD) Type [Count of Participants; unit: Participants] — Hemoglobin SS disease is the most common type of sickle cell disease and the most severe form of SCD. Hemoglobin SC disease is the second most common type of sickle cell disease. Symptoms are similar to individuals with Hb SS, but the anemia is less severe.
  Participants
    SS | 9
    SC | 7
    Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of VR Session as Measured by Patient Satisfaction Survey.
Description: Patient satisfaction with session measured on a Likert-type scale with the following options: Very unsatisfied, unsatisfied, not unsatisfied or satisfied, satisfied, very satisfied. Participants were also asked if they agree with the statement that the 'VR device was helpful'.
Time Frame: Day 1
Population: Data not collected on 8 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | VR Intervention Session
Number analyzed (Participants) | 12
Participants
  'Satisfied' to 'very satisfied' | 9
  Agree with the statement that the 'VR device was helpful' | 11

2. Secondary Outcome: Change in Pain Score
Description: Change in pain score as measured by visual analog pain score (0-10), where 0 = no pain and 10 = worst pain.
Time Frame: Baseline, up to 30 mins
Population: Three participants did not have both a before and an after score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR Intervention Session
Number analyzed (Participants) | 17
score on a scale | -0.88 (0.53)
Statistical Analysis 1: Comparison: VR Intervention Session; Test type: Other; p < 0.005, Paired t-test

3. Secondary Outcome: Change in Anxiety-related Symptoms as Measured by Generalized Anxiety Disorder-7 (GAD-7) Score
Description: GAD-7 total score for the seven items ranges from 0 to 21, calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." A total score of 0-4 = minimal anxiety, 5-9 = mild anxiety, 10-14 = moderate anxiety, 15-21 = severe anxiety. A negative score change indicates a decrease in anxiety symptoms and a positive score change indicates an increase in anxiety symptoms.
Time Frame: Baseline, up to 30 mins
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR Intervention Session
Number analyzed (Participants) | 20
score on a scale | -1.80 (1.62)
Statistical Analysis 1: Comparison: VR Intervention Session; Test type: Other; p < 0.05, Paired t-test

4. Secondary Outcome: Change in Depressive Symptoms as Measured by Patient Health Questionnaire-9 (PHQ-9) Score
Description: The PHQ-9 has a total range of 0-27, where 0 = No depression, 1-4 = Minimal depression, 5-9 = Mild depression, 10-14 = Moderate depression, 15-19 = Moderately severe depression, 20-27 = Severe depression. A negative score change indicates a decrease in depressive symptoms and a positive score change indicates an increase in depressive symptoms.
Time Frame: Baseline, up to 30 mins
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR Intervention Session
Number analyzed (Participants) | 20
score on a scale | -1.85 (1.57)
Statistical Analysis 1: Comparison: VR Intervention Session; Test type: Other; p < 0.05, Paired t-test

ADVERSE EVENTS:
Time Frame: During virtual reality (VR) session, up to 30 minutes
Arm/Group | VR Intervention Session
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT03387033/Prot_SAP_000.pdf